CLINICAL TRIAL: NCT02186561
Title: Prospective Study on Embolization of Intracranial Aneurysms With the Pipeline™ Device (PREMIER)
Brief Title: Prospective Study on Embolization of Intracranial Aneurysms With Pipeline™ Embolization Device
Acronym: PREMIER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Neurovascular Clinical Affairs (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NV-PED-07; NCT02178007 (obsolete NCT alias)
Record Dates: First submitted 2014-07-08; First posted 2014-07-10 (Estimated); Results first posted 2019-05-21 (Actual); Last update posted 2019-12-27 (Actual); Status verified 2019-12

CONDITIONS: Intracranial Aneurysm
Keywords: Intracranial aneurysm; brain aneurysm
MeSH Terms: conditions — Intracranial Aneurysm

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Device: Yes

ARMS (1):
- Pipeline™ Embolization Device (Experimental): treatment with Pipeline™ Embolization Device
  Interventions: Device: Pipeline™ Embolization Device/ Pipeline™Flex Embolization Device

INTERVENTIONS:
Device: Pipeline™ Embolization Device/ Pipeline™Flex Embolization Device

SUMMARY:
The purpose of this study is to assess the safety and effectiveness of the Pipeline™ device in the treatment of unruptured, wide-neck intracranial aneurysms.

ELIGIBILITY:
Inclusion Criteria:

1. Subject has provided written informed consent using the IRB/EC-approved consent form and agrees to comply with protocol requirements.
2. Age 22-80 years.
3. Subject has a target intracranial aneurysm (IA) located in the:

   1. Internal carotid artery (up to the carotid terminus) OR
   2. Vertebral artery segment up to and including the posterior inferior cerebellar artery
4. Subject has a target IA that is ≤ 12 mm.
5. Subject has a target IA that has a parent vessel with diameter 1.5-5.0 mm distal/proximal to the target IA.
6. Subject has a target IA with an aneurysm neck ≥ 4mm or a dome to neck ratio ≤ 1.5.
7. Subject has a pre-procedure PRU value between 60-200.

Exclusion Criteria:

1. Subject has received an intracranial implant (e.g. coils) in the area of the target IA within the past 12 weeks.
2. Subarachnoid hemorrhage in the past 30 days.
3. Subject with anatomy not appropriate for endovascular treatment due to severe intracranial vessel tortuosity or stenosis determined from baseline or pre-procedure imaging, or a history of intracranial vasospasm not responsive to medical therapy.
4. Major surgery in the last 30 days.
5. History of irreversible bleeding disorder and/or subject presents with signs of active bleeding.
6. Any known contraindication to treatment with the Pipeline™ device, including:

   1. Stent is in place in the parent artery at the target IA location
   2. Contraindication to dual antiplatelet therapy
   3. Relative contraindication to angiography (e.g., serum creatinine >2.5 mg/dL, allergy to contrast that cannot be medically controlled).
   4. Known severe allergy to platinum or cobalt/chromium alloys.
   5. Evidence of active infection at the time of treatment (e.g., fever with temperature >38°C and/or WBC >1.5 109/L).
7. The Investigator determines that the health of the subject or the validity of the study outcomes (e.g., high risk of neurologic events, worsening of clinical condition in the last 30 days) may be compromised by the subject's enrollment.
8. Pregnant or breast-feeding women or women who wish to become pregnant during the length of study participation.
9. Participating in another clinical trial during the follow-up period that could confound the treatment or outcomes of this investigation.

Ages: 22 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 197 (Actual)
Dates: Start 2014-07-24 (Actual); Primary Completion 2016-11-18 (Actual); Study Completion 2018-12-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ricardo Hanel, M.D., Principal Investigator — Baptist Medical Center
Locations (23):
- United States (22):
  - Radiology Imaging Associates, Englewood, Colorado
  - Baptist Medical Center Jacksonville, Jacksonville, Florida
  - Tampa General Hospital, Tampa, Florida
  - Florida Hospital, Winter Park, Florida
  - The Emory Clinic, Atlanta, Georgia
  - Rush University Medical Center, Chicago, Illinois
  - Baptist Physicians Lexington, Lexington, Kentucky
  - University of Kentucky, Lexington, Kentucky
  - The Johns Hopkins Hospital, Baltimore, Maryland
  - Tufts University Medical Center, Boston, Massachusetts
  - University of Massachusetts Memorial Medical Center, Worcester, Massachusetts
  - Mayo Clinic Rochester, Rochester, Minnesota
  - Kaleida Health/University of Buffalo, Buffalo, New York
  - Stony Brook University, Stony Brook, New York
  - Cleveland Clinic, Cleveland, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - Geisinger Medical Center, Danville, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - St. Luke's Health Baylor College of Medicine, Houston, Texas
  - The Methodist Hospital, Houston, Texas
  - University of Utah, Salt Lake City, Utah
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin
- Toronto Western Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
No, there is not a plan to make IPD available.

REFERENCES:
- [Derived] Rodriguez-Erazu F, Cortez GM, Lopes DK, Gutierrez-Aguirre SF, De Toledo OF, Aghaebrahim A, Sauvageau E, Kallmes DF, Fiehler J, Hanel RA. Braids and beyond: a comprehensive study on pipeline device braid stability from PREMIER data. J Neurointerv Surg. 2025 Nov 18;17(12):1362-1367. doi: 10.1136/jnis-2024-022350. PMID 39357888
- [Derived] Hanel RA, Cortez GM, Lopes DK, Nelson PK, Siddiqui AH, Jabbour P, Mendes Pereira V, Istvan IS, Zaidat OO, Bettegowda C, Colby GP, Mokin M, Schirmer CM, Hellinger FR, Given C, Krings T, Taussky P, Toth G, Fraser JF, Chen M, Priest R, Kan P, Fiorella D, Frei D, Aagaard-Kienitz B, Diaz O, Malek AM, Cawley CM, Puri AS, Kallmes DF. Prospective study on embolization of intracranial aneurysms with the pipeline device (PREMIER study): 3-year results with the application of a flow diverter specific occlusion classification. J Neurointerv Surg. 2023 Mar;15(3):248-254. doi: 10.1136/neurintsurg-2021-018501. Epub 2022 Mar 15. PMID 35292570
- [Derived] Hanel RA, Kallmes DF, Lopes DK, Nelson PK, Siddiqui A, Jabbour P, Pereira VM, Szikora Istvan I, Zaidat OO, Bettegowda C, Colby GP, Mokin M, Schirmer C, Hellinger FR, Given Ii C, Krings T, Taussky P, Toth G, Fraser JF, Chen M, Priest R, Kan P, Fiorella D, Frei D, Aagaard-Kienitz B, Diaz O, Malek AM, Cawley CM, Puri AS. Prospective study on embolization of intracranial aneurysms with the pipeline device: the PREMIER study 1 year results. J Neurointerv Surg. 2020 Jan;12(1):62-66. doi: 10.1136/neurintsurg-2019-015091. Epub 2019 Jul 15. PMID 31308197

RESULTS

PARTICIPANT FLOW:
Groups:
- PREMIER: The investigational device was implanted in the internal carotid artery (up to the terminus) or the vertebral artery segment up to and including the posterior inferior cerebellar artery to treat unruptured, wide-necked, aneurysms measuring ≤ 12 mm.
Period: Enrollment
Arm/Group | PREMIER
Started (Participants Consented and Assessed for Eligibility) | 197
Completed (Enrolled Participants in Whom Deployment of the Investigational Device was Attempted- ITT Population) | 141
Not Completed | 56
Not completed — Did Not Meet Inclusion Criteria | 46
Not completed — Enrollment Cap Reached | 5
Not completed — Insurance Denial | 2
Not completed — Withdrawal by Subject | 2
Not completed — Investigator Withdrew Consent | 1
Period: Subjects Implanted With Device
Arm/Group | PREMIER
Started (Participants with an Attempted Investigational Device Implant) | 141
Completed (Participants with a Successful Investigational Device Implant) | 141
Not Completed | 0
Period: 30-Day Post Index Procedure Visit
Arm/Group | PREMIER
Started (Participants implanted with the investigational device.) | 141
Completed (Participants Implanted with the Investigational Device that Completed the 30 Day Visit) | 140
Not Completed | 1
Not completed — Death | 1
Period: 180- Day Post Index Procedure Visit
Arm/Group | PREMIER
Started (Participants implanted with the investigational device.) | 141
Completed (Participants Implanted with the Investigational Device that Completed the 30 Day Visit) | 134
Not Completed | 7
Period: 1- Year Post Index Procedure Visit
Arm/Group | PREMIER
Started (Participants implanted with the investigational device.) | 141
Completed (Participants Implanted with the Investigational Device that Completed the 1 Year Visit) | 139
Not Completed | 2
Not completed — Death | 1
Not completed — Missed | 1
Period: 2 - Year Post Index Procedure Visit
Arm/Group | PREMIER
Started (Participants implanted with the investigational device.) | 141
Completed (Participants Implanted with the Investigational Device that Completed the 2 Year Visit) | 134
Not Completed | 7
Period: 3 - Year Post Index Procedure Visit
Arm/Group | PREMIER
Started (Participants implanted with the investigational device.) | 141
Completed (Participants Implanted with the Investigational Device that Completed the 3 Year Visit) | 128
Not Completed | 13

BASELINE CHARACTERISTICS:
Population: Intent to Treat Population was defined as all enrolled participants in whom deployment of the Investigational device was attempted.
Arm/Group | PREMIER
Number analyzed (Participants) | 141
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.6 (11.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 124
  Male | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 12
  Not Hispanic or Latino | 115
  Unknown or Not Reported | 14
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 4
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 16
  White | 114
  More than one race | 0
  Unknown or Not Reported | 6
Region of Enrollment [Number; unit: participants]
  Canada | 6
  United States | 135

OUTCOME MEASURES:

1. Primary Outcome: The Percentage of Participants With the Occurrence of Major Stroke in the Territory Supplied by the Treated Artery or Neurological Death at 12-Months Post Procedure
Description: The primary safety endpoint was defined as a stroke which results in focal neurological deficit for 24 hrs or more and increases the NIH Stroke Scale of the subject by ≥ 4 along with an imaging correlate. Missing data for subjects who failed to complete the 12- month post-procedure evaluation without any evidence of a major stroke in the territory supplied by the treated artery or neurological death were imputed in the analysis using multiple imputation. Multiple imputation provides a mechanism for deriving estimates for a population where not all of the patients have an endpoint determination.
Time Frame: Up to 12 Months Post Procedure
Population: Participants enrolled and implanted with the Investigational Device (ITT)
Measure: Number; unit: percentage of participants
Arm/Group | PREMIER
Number analyzed (Participants) | 141
percentage of participants | 2.17

2. Primary Outcome: The Percentage of Participants With Complete Aneurysm Occlusion (Defined as Raymond Roy Grade 1) Without Significant Parent Artery Stenosis (≤ 50%) or Retreatment of the Target Aneurysm at 12-Months Post-Procedure
Description: The definitions for the three components of the primary effectiveness endpoint were: 1) retreatment, defined as all retreatment procedures occurring between the index procedure and 1 Year post-procedure; 2) complete aneurysm occlusion based on Core Laboratory review of 1-year images and 3) significant parent artery stenosis, based on Core Laboratory review of 1-year images. The Raymond-Roy Grading scale is used for judging intracranial aneurysm (IA) endosaccular embolization success. Grade I is completion occlusion with no flow of contrast seen in the aneurysm sac, Grade II is partial occlusion with some flow or eddy flow in the aneurysm sac and Grade III is residual aneurysm or Incomplete occlusion with apparent flow in the aneurysm sac.
  Multiple imputation provides a mechanism for deriving estimates for a population where not all of the patients have an endpoint determination.
Time Frame: Up to 12 Months Post Procedure
Population: Participants Treated with Investigational Device that Completed the 12 Month Visit Imaging
Measure: Number; unit: Percentage of Participants
Arm/Group | PREMIER
Number analyzed (Participants) | 141
Percentage of Participants | 76.71

3. Secondary Outcome: The Number of Participants With a Major Stroke in the Territory Supplied by the Treated Artery or Neurological Death at 30-days Post Procedure Due to Procedural Complications
Description: Major Stroke is defined as a stroke which results in focal neurological deficit for 24 hrs or more and increases the NIH Stroke Scale of the subject by ≥ 4 along with an imaging correlate. Neurological death is any subject death due to neurologic reasons.
Time Frame: Up to 30 days, Post Procedure
Population: Participants Treated with the Investigational Device that Completed the 30 Day Visit
Measure: Count of Participants; unit: Participants
Arm/Group | PREMIER
Number analyzed (Participants) | 141
Participants | 0

4. Secondary Outcome: The Number of Participants Who Experienced Delayed Intracerebral Hemorrhage > 30 Days Post-Procedure
Description: For the purpose of this protocol, delayed intracerebral hemorrhage was defined as hemorrhage within the fixed vault of the cranium (skull) occurring greater than 30 days post-procedure.
Time Frame: > 30 days, Post Procedure
Population: ParticipantsTreated with the Investigational Device that Completed the 30 Day Visit
Measure: Number; unit: Participants
Arm/Group | PREMIER
Number analyzed (Participants) | 141
Participants | 1

5. Secondary Outcome: The Number of Participants With Successfully Deployed Investigational Device
Description: The secondary outcome measures provides the number of participants successfully implanted with the Investigational device during the study index procedure at the target site.
Time Frame: Index Procedure
Population: Participants Enrolled who Underwent the Index Procedure
Measure: Count of Participants; unit: Participants
Arm/Group | PREMIER
Number analyzed (Participants) | 141
Participants | 140

ADVERSE EVENTS:
Time Frame: Adverse Events were collected from the point of consent through year 3
Description: The adverse event data reported by sites was adjudicated by a three member independent Clinical Events Committee (CEC). All data presented within this section has been CEC adjudicated.
  Adjudicable events met the following criteria:
  * All Adverse Events (AE) with an underlying neurological cause (Neurological Adverse Events)
  * All Device Related Adverse Events
  * All Procedure Related Adverse Events
  * All Serious Adverse Events (SAE's)
Groups:
- CEC Adjudicated Adverse Events Through 1-Year: Participants who received the Investigational Device followed through 1 Year
- CEC Adjudicated Adverse Events Through 2-Year: Participants who received the Investigational Device followed through 2 Year
- CEC Adjudicated Adverse Events Through 3-Year: Participants who received the Investigational Device followed through 3 Year
Arm/Group | CEC Adjudicated Adverse Events Through 1-Year | CEC Adjudicated Adverse Events Through 2-Year | CEC Adjudicated Adverse Events Through 3-Year
All-Cause Mortality (participants affected / at risk) | 1/141 | 1/141 | 2/141
Serious Adverse Events (participants affected / at risk) | 39/141 | 49/141 | 60/141
Other Adverse Events (participants affected / at risk) | 107/141 | 112/141 | 112/141
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CEC Adjudicated Adverse Events Through 1-Year (N=141) | CEC Adjudicated Adverse Events Through 2-Year (N=141) | CEC Adjudicated Adverse Events Through 3-Year (N=141)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 1 (2)
Atrial flutter (Cardiac disorders) | 1 (1) | 1 (1) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 1 (1) | 1 (1)
Coronary Artery Disease (Cardiac disorders) | 0 (0) | 2 (2) | 3 (3)
Ventricular tachycardia (Cardiac disorders) | 1 (1) | 1 (1) | 1 (1)
Vision Blurred (Eye disorders) | 1 (1) | 1 (1) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 3 (5) | 3 (5) | 3 (5)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1)
Peritoneal haemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1)
Adverse drug reaction (General disorders) | 2 (2) | 2 (2) | 2 (2)
Chest pain (General disorders) | 1 (1) | 2 (3) | 3 (4)
Thrombosis in Device (General disorders) | 1 (1) | 1 (1) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 2 (2)
Portal vein thrombosis (Hepatobiliary disorders) | 1 (1) | 1 (1) | 1 (1)
Anaphylactic reaction (Immune system disorders) | 1 (1) | 1 (1) | 1 (1)
Colonic abscess (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Diverticulitis (Infections and infestations) | 1 (1) | 1 (1) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1) | 1 (1) | 1 (1)
Influenza (Infections and infestations) | 1 (1) | 1 (1) | 2 (2)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Upper Respiratory Tract Infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Wound Infection (Infections and infestations) | 1 (1) | 1 (1) | 1 (1)
Patella Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1)
Procedural hypertension (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 1 (1)
Vascular Graft Occlusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1)
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 1 (2) | 1 (2) | 1 (2)
Back Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Compartment syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 1 (1)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 1 (1)
Basal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 1 (1)
Carotid Artery Dissection (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1)
Carotid artery stenosis (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1)
Cerebral Haemorrhage (Nervous system disorders) | 3 (3) | 4 (4) | 4 (4)
Cerebral Infarction (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1)
Convulsion (Nervous system disorders) | 0 (0) | 3 (3) | 3 (3)
Headache (Nervous system disorders) | 4 (5) | 5 (6) | 6 (7)
Ischaemic stroke (Nervous system disorders) | 3 (4) | 3 (4) | 3 (4)
Migraine (Nervous system disorders) | 2 (2) | 3 (3) | 3 (3)
Multiple sclerosis relapse (Nervous system disorders) | 1 (1) | 1 (1) | 1 (2)
Myasthenia Gravis (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Presyncope (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 2 (2) | 3 (3)
Delirium (Psychiatric disorders) | 1 (1) | 1 (1) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 1 (1) | 2 (2)
Major depression (Psychiatric disorders) | 1 (1) | 1 (1) | 1 (2)
Suicide Attempt (Psychiatric disorders) | 1 (1) | 1 (1) | 2 (2)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1)
Renal failure chronic (Renal and urinary disorders) | 1 (1) | 1 (1) | 1 (1)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 (1) | 1 (1) | 1 (1)
Ovarian cyst ruptured (Reproductive system and breast disorders) | 1 (1) | 1 (1) | 1 (1)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 2 (2)
Stevens-Johnson Syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Aneurysm repair (Surgical and medical procedures) | 5 (5) | 9 (9) | 9 (9)
Haematoma (Vascular disorders) | 1 (1) | 1 (1) | 1 (1)
Hypertensive Crisis (Vascular disorders) | 1 (1) | 3 (3) | 3 (5)
Vascular Occlusion (Vascular disorders) | 1 (1) | 1 (1) | 1 (1)
Lymphatic Disorder (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (2)
Cardiac Arrest (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Gastritis Erosive (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Bronchopulmonary Aspergillosis Allergic (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Overdose (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (2)
Tibia Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Loss of Consciousness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Suicidal Ideation (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Menorrhagia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Ovarian Cyst (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (2)
Coronary Arterial Stent Insertion (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Intervertebral Disc Operation (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Medical Device Removal (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Malignant Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Vascular Occlusion (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CEC Adjudicated Adverse Events Through 1-Year (N=141) | CEC Adjudicated Adverse Events Through 2-Year (N=141) | CEC Adjudicated Adverse Events Through 3-Year (N=141)
Haemorrhagic Diathesis (Blood and lymphatic system disorders) | 2 (2) | 2 (2) | 2 (2)
Lymphoid tissue hyperplasia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 2 (2) | 2 (2) | 2 (2)
Vertigo positional (Ear and labyrinth disorders) | 1 (1) | 1 (1) | 1 (1)
Amaurosis Fugax (Eye disorders) | 0 (0) | 1 (1) | 1 (1)
Blepharospasm (Eye disorders) | 1 (1) | 2 (2) | 2 (2)
Conjunctival Haemorrhage (Eye disorders) | 1 (1) | 1 (1) | 1 (1)
Diplopia (Eye disorders) | 3 (3) | 3 (3) | 3 (3)
Eye pain (Eye disorders) | 2 (2) | 2 (2) | 2 (2)
Photophobia (Eye disorders) | 1 (2) | 2 (3) | 2 (3)
Photopsia (Eye disorders) | 2 (2) | 2 (2) | 2 (2)
Vision blurred (Eye disorders) | 7 (7) | 8 (8) | 8 (8)
Visual impairment (Eye disorders) | 15 (15) | 17 (17) | 17 (17)
Vitreous detachment (Eye disorders) | 1 (1) | 1 (1) | 1 (1)
Vitreous floaters (Eye disorders) | 5 (5) | 5 (5) | 5 (5)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Gastrointestinal inflammation (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1)
Hiatus hernia (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1)
Nausea (Gastrointestinal disorders) | 3 (3) | 3 (3) | 3 (3)
Adverse drug reaction (General disorders) | 1 (1) | 1 (1) | 1 (1)
Catheter site haematoma (General disorders) | 13 (13) | 13 (13) | 13 (13)
Catheter site haemorrhage (General disorders) | 9 (9) | 9 (9) | 9 (9)
Catheter site pain (General disorders) | 6 (6) | 6 (6) | 6 (6)
Fatigue (General disorders) | 1 (1) | 1 (1) | 1 (1)
Local swelling (General disorders) | 1 (1) | 1 (1) | 1 (1)
Catheter site infection (Infections and infestations) | 1 (1) | 1 (1) | 1 (1)
Concussion (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 1 (1)
Periorbital Haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 1 (1)
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 1 (1)
Hypervolaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 1 (1)
Hypovolaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 1 (1)
Spinal Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 1 (1)
Aphasia (Nervous system disorders) | 3 (3) | 4 (4) | 4 (4)
Ataxia (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Balance disorder (Nervous system disorders) | 3 (3) | 3 (3) | 3 (3)
Carpal Tunnel Syndrome (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Cerebral infarction (Nervous system disorders) | 2 (2) | 2 (2) | 2 (2)
Cerebral vasoconstriction (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1)
Convulsion (Nervous system disorders) | 0 (0) | 1 (1) | 2 (2)
Disturbance in attention (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1)
Dizziness (Nervous system disorders) | 5 (6) | 9 (11) | 9 (12)
Dysarthria (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Haemorrhage intracranial (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1)
Headache (Nervous system disorders) | 33 (35) | 34 (38) | 38 (44)
Hemiparesis (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 2 (2) | 2 (2) | 2 (2)
Intracranial Artery Dissection (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1)
Ischaemic Stroke (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1)
Migraine (Nervous system disorders) | 2 (2) | 2 (2) | 2 (2)
Muscle spasticity (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1)
Neuropathy peripheral (Nervous system disorders) | 2 (2) | 2 (2) | 2 (2)
Paraesthesia (Nervous system disorders) | 5 (5) | 6 (6) | 7 (7)
Presyncope (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1)
Radiculitis Lumbosacral (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Radiculopathy (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Sensory Disturbance (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1)
Subarachnoid Heamorrhage (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1)
Syncope (Nervous system disorders) | 3 (3) | 4 (4) | 4 (4)
Transient Ischaemic Attack (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1)
Tremor (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1)
Visual field defect (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1)
Confusional state (Psychiatric disorders) | 1 (1) | 1 (1) | 1 (1)
Dysphemia (Psychiatric disorders) | 1 (1) | 1 (1) | 1 (1)
Mental status changes (Psychiatric disorders) | 1 (1) | 1 (1) | 1 (1)
Menorrhagia (Reproductive system and breast disorders) | 1 (1) | 1 (1) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 4 (4) | 4 (4)
Alopecia (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2) | 2 (2)
Ecchymosis (Skin and subcutaneous tissue disorders) | 28 (28) | 29 (29) | 29 (29)
Petechiae (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 1 (1)
Swelling Face (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 1 (1)
Arterial stenosis (Vascular disorders) | 4 (4) | 4 (4) | 6 (6)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 1 (1) | 1 (1)
Flushing (Vascular disorders) | 1 (1) | 1 (1) | 1 (1)
Haematoma (Vascular disorders) | 1 (1) | 1 (1) | 1 (1)
Haemorrhage (Vascular disorders) | 1 (1) | 1 (1) | 1 (1)
Hypotension (Vascular disorders) | 1 (1) | 1 (1) | 1 (1)
Vasospasm (Vascular disorders) | 28 (29) | 28 (29) | 29 (31)
Catheter Site Injury (General disorders) | 0 (0) | 0 (0) | 1 (1)
Modified Rankin Score Decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Back Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Cognitive Disorder (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Monoplegia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Deep Vein Thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-03-24): https://cdn.clinicaltrials.gov/large-docs/61/NCT02186561/Prot_SAP_000.pdf